CLINICAL TRIAL: NCT02820129
Title: Effectiveness of a Medication Wallet Card
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TAPER-Wallet-Card-002-May-23
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Comorbidity; Medication Therapy Management; Polypharmacy
Keywords: polypharmacy; wallet card; medication; self-efficacy; patient enablement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wallet Card Group (Experimental): The intervention arm is comprised of:
  Patients from the TAPER study who receive a medication wallet card with their medications and medical conditions listed.
  Interventions: Device: Medication Wallet Card
- Control Group (Placebo Comparator): Standard of care as well as wait list control. These participants will receive a "reminder" wallet card which states, "Remember to keep an up-to-date listing of your medications and bring your medications to your doctor's appointments."
  Interventions: Device: Reminder Card

INTERVENTIONS:
Device: Medication Wallet Card — A medication wallet card will be given to the intervention group. This will be personalized for each patient and will include the patient's medications, dosages, and medical conditions. It will be personally given to a patient after a medical appointment with their family physician.
  Arms: Wallet Card Group
Device: Reminder Card — A reminder card will be given to this group. The card will not be personal and will be mailed to patients. It will state, "Remember to keep an up-to-date listing of your medications and bring your medications to your doctor's appointments."
  Other Names: Placebo Intervention
  Arms: Control Group

SUMMARY:
This study evaluates whether or not the use of a medication wallet card in patients over 70 taking 5 or more medications promotes self-efficacy with regards to coping with illness, understanding medications, and staying healthy. Half of the participants will receive an individualized medication wallet card with their medications and medical conditions listed while the other half will receive a simple reminder card.

DETAILED DESCRIPTION:
In order to prevent medication errors and subsequent ADEs, a complete and accurate medication list must be maintained. Although electronic healthcare records, maintained by healthcare providers, have been praised for their potential to decrease medication errors, studies show that the sole implementation of a paperless system is not sufficient to eliminate medication recording and prescription errors. Hence, an approach to maintain complete medication lists will need to involve the cooperation of both health care providers and patients. A previous study showed that an integrated approach including all members of the healthcare team and the patient improved the completeness and accuracy of medication list from 7.7% to 18.5%. One way to increase patient involvement in medication reconciliation is by allowing the patients to become more informed about their health and medications.

According to the Bandura's Social Cognitive Theory of Self-Efficacy, the beliefs a person holds regarding his or her power to influence situations strongly affects the agency a person has to face challenges capably. A tool such as an up-to-date MWC that has a list of the medications and dosages in addition to medical conditions listed may help older patients to better understand and manage their health. Furthermore, a wallet card has been an effective tool with many benefits. For example, a study showed that a Medication Allergy Profile card increased patient's knowledge of their drug regimens, decreased medication errors, decreased drug interactions, and improved patients' compliance.

No randomized control trials currently show the the impact of a medication wallet card/list on patient enablement. One study showed that a significant percentage of the patients were willing to use a self-maintained wallet-sized medication list. In addition, those who used the medication list showed an improved sense of knowledge about their medical problems and medication, and also exhibited an enhanced sense of responsibility in maintaining their medication lists. However, the study considered a relatively young population that only included patients over the age of 40 and did not stipulate a minimum number of medications for the patients to be taking. In addition, the study was not a randomized control trial, and used the Patient Medication Scale (PMS) to measure outcomes.

Hence, a randomized control trial employing a standardized questionnaires to investigate an older population (age greater than 70) experiencing polypharmacy is needed to asses the impact of a medical wallet card in promoting self efficacy and patient enablement.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years of age or older
* Participating family doctor as most responsible provider
* Patient of McMaster Family Health Team
* Currently taking 5 or more medications
* Have not had a recent comprehensive medication review
* Patient consents

Exclusion Criteria:

* English language or cognitive skills inadequate to understand and respond to rating scales
* Terminal illness or other circumstance precluding 13 month study period

Ages: 70 Years to 116 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient Enablement Index | 4 weeks
  Patient Enablement Index
Patient Enablement Index | 6 months
  Patient Enablement Index Repeated

SECONDARY OUTCOMES:
Usability - Qualitative Data | 4 weeks
  Survey questions by telephone assessing the usability of a medication wallet card. Questions include: How clear was your medication wallet card? How did you use your medication wallet card over the past four weeks? Did your medication wallet card help you over the past four weeks? If so, how? Do you intend on continuing to carry your medication wallet card?

CONTACTS AND LOCATIONS:
Overall Officials: Ainsley Moore, MD, Principal Investigator — McMaster University, Department of Family Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillestad R, Bigelow J, Bower A, Girosi F, Meili R, Scoville R, Taylor R. Can electronic medical record systems transform health care? Potential health benefits, savings, and costs. Health Aff (Millwood). 2005 Sep-Oct;24(5):1103-17. doi: 10.1377/hlthaff.24.5.1103. PMID 16162551
- [Background] Varkey P, Cunningham J, Bisping DS. Improving medication reconciliation in the outpatient setting. Jt Comm J Qual Patient Saf. 2007 May;33(5):286-92. doi: 10.1016/s1553-7250(07)33033-x. PMID 17503684
- [Background] Nassaralla CL, Naessens JM, Chaudhry R, Hansen MA, Scheitel SM. Implementation of a medication reconciliation process in an ambulatory internal medicine clinic. Qual Saf Health Care. 2007 Apr;16(2):90-4. doi: 10.1136/qshc.2006.021113. PMID 17403752
- [Background] Gandhi TK, Weingart SN, Seger AC, Borus J, Burdick E, Poon EG, Leape LL, Bates DW. Outpatient prescribing errors and the impact of computerized prescribing. J Gen Intern Med. 2005 Sep;20(9):837-41. doi: 10.1111/j.1525-1497.2005.0194.x. PMID 16117752
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Klein GL, Zenk KE. A Medical Allergy Profile (MAP) card. Ann Allergy. 1981 Jun;46(6):328-30. PMID 7247083
- [Background] Chae SY, Chae MH, Isaacson N, James TS. The patient medication list: can we get patients more involved in their medical care? J Am Board Fam Med. 2009 Nov-Dec;22(6):677-85. doi: 10.3122/jabfm.2009.06.090059. PMID 19897697
- [Background] Hudon C, Fortin M, Rossignol F, Bernier S, Poitras ME. The Patient Enablement Instrument-French version in a family practice setting: a reliability study. BMC Fam Pract. 2011 Jul 7;12:71. doi: 10.1186/1471-2296-12-71. PMID 21736729